CLINICAL TRIAL: NCT04610827
Title: Optimum Frequency and Timing of Oral Iron Administration for Childhood Restless Leg Syndrome/Periodic Limb Movement Disorder
Brief Title: Oral Iron Frequency for Childhood Restless Leg Syndrome/Periodic Limb Movement Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Change in personnel and lack of resources to continue.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Julie M. Baughn, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-007655
Record Dates: First submitted 2020-10-26; First posted 2020-11-02 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Sleep Disorder; Restless Legs Syndrome; Periodic Limb Movement Sleep Disorder; Iron-deficiency
MeSH Terms: conditions — Sleep Wake Disorders; Restless Legs Syndrome; Anemia, Iron-Deficiency | interventions — ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ferrous sulfate daily (Active Comparator): Subject will take 3 mg/kg oral iron in the morning
  Interventions: Drug: Ferrous sulfate
- Ferrous sulfate twice daily (Active Comparator): Subjects will take 1.5 mg/kg oral iron twice daily
  Interventions: Drug: Ferrous sulfate
- Ferrous sulfate every other day (Active Comparator): 6 mg/kg oral iron every other day in the morning
  Interventions: Drug: Ferrous sulfate

INTERVENTIONS:
Drug: Ferrous sulfate — Guideline-recommended 3 mg/kg/day dosing

SUMMARY:
The purpose of this research study is to see if the level of serum ferritin differs based on how often oral iron (in the form of ferrous sulfate) is given to children with restless leg syndrome/periodic limb movement disorder.

ELIGIBILITY:
Inclusion Criteria:

* Ferritin equal to or lower than 24 mcg/L drawn within the last 30 days.
* Age 2 to 10 years.
* Diagnosis of restless leg syndrome, periodic limb movement disorder, or sleep disturbance.

Exclusion Criteria:

* Currently taking oral formulation of iron other than a multivitamin.
* Untreated obstructive sleep apnea.
* Gastrointestinal disorder, including gastroesophageal reflux disease and celiac disease.
* Prior gastrointestinal surgery; e.g., gastrectomy, duodenal bypass, and presence of G-tube.
* Use of H2 blocker, antacid, or proton pump inhibitor.
* Inflammatory disorders, including juvenile idiopathic arthritis or inflammatory bowel disease.
* Elevated CRP at time of initial ferritin or report of illness in past 4 weeks.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Baughn, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ferrous Sulfate Daily | Ferrous Sulfate Twice Daily | Ferrous Sulfate Every Other Day
Started | 1 | 2 | 3
Completed | 0 | 1 | 3
Not Completed | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferrous Sulfate Daily | Ferrous Sulfate Twice Daily | Ferrous Sulfate Every Other Day | Total
Number analyzed (Participants) | 1 | 2 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 3 | 6
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2
  Male | 0 | 1 | 3 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Ferritin Level
Description: Ferritin level in blood measured in micrograms per liter
Time Frame: 2 months
Population: Ferritin level at 2 months was not collected for 4 participants.
Measure: Number; unit: mcg/L
Arm/Group | Ferrous Sulfate Daily | Ferrous Sulfate Twice Daily | Ferrous Sulfate Every Other Day
Number analyzed (Participants) | 0 | 1 | 1
mcg/L |  | 24 | 19

2. Primary Outcome: Side Effects
Description: Number of subjects to experience side effects effects (e.g., stool color change, nausea, constipation, teeth staining)
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ferrous Sulfate Daily | Ferrous Sulfate Twice Daily | Ferrous Sulfate Every Other Day
Number analyzed (Participants) | 1 | 2 | 3
Participants | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 2 months after starting ferrous sulfate on all participants.
Arm/Group | Ferrous Sulfate Daily | Ferrous Sulfate Twice Daily | Ferrous Sulfate Every Other Day
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 1/1 | 1/2 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferrous Sulfate Daily (N=1) | Ferrous Sulfate Twice Daily (N=2) | Ferrous Sulfate Every Other Day (N=3)
Nausea/GI Upset (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study terminated due to change in personnel and lack of resources to continue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT04610827/Prot_SAP_000.pdf